CLINICAL TRIAL: NCT07051824
Title: The Effect of Probiotic and Prebiotic Use on Gastrointestinal System and Some Biochemical Parameters in the Early Postoperative Period of Sleeve Gastrectomy Patients
Brief Title: Probiotic and Prebiotic Use in Early Postoperative Period of Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayten Altunsaray (Other Government)
Responsible Party: Sponsor-Investigator, Ayten Altunsaray, Principal Investigator, Lokman Hekim University
Organization: Lokman Hekim University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240239
Record Dates: First submitted 2025-06-17; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Sleeve Gastrectomy; Gastrointestinal Symptoms; Prebiotic; Probiotic
Keywords: Gastrointestinal Symptoms; Prebiotic; Probiotic; Sleeve Gastrectomy
MeSH Terms: interventions — Probiotics; Prebiotics; maltodextrin; guar gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Probiotic and Prebiotic) (Experimental): Participants received a daily 5 g sachet containing:
  * Partially hydrolyzed guar gum (PHGG): 4.9 g (prebiotic fiber),
  * Lactobacillus rhamnosus GG (LGG): 1×10⁹ CFU (probiotic),
  * Maltodextrin: 0.1 g (excipient).
  The sachet was mixed with 200 ml yogurt and consumed as an afternoon snack for 12 weeks post-surgery.
  Interventions: Dietary Supplement: Probiotic and Prebiotic
- Control Group (No intervention) (No Intervention): Standard Care Control Participants followed routine post-operative care without dietary supplements.

INTERVENTIONS:
Dietary Supplement: Probiotic and Prebiotic — This synbiotic intervention aims to minimize postoperative gastrointestinal symptoms in sleeve gastrectomy patients. The 5 g sachet contains:
  * Partially hydrolyzed guar gum (PHGG; 4.9 g): Clinically shown to reduce diarrhea and improve stool consistency,
  * Lactobacillus rhamnosus GG (LGG; 1×10⁹ CFU): Evidence-based for alleviating abdominal pain and bloating,
  * Maltodextrin (0.1 g): Excipient for stability.
  Administered daily in yogurt for 12 weeks post-surgery, this combination directly targets:
  ① Diarrhea and constipation (via PHGG's soluble fiber),
  ② Abdominal pain and bloating (via LGG's anti-inflammatory effects),
  ③ Overall GI symptom burden.
  **Distinctive features vs. other studies:
  * Symptom-specific formulation: PHGG (high-dose fiber) + LGG (symptom-targeted probiotic) synergy,
  * Surgical context: Optimized for rapid gastric transit post-sleeve gastrectomy,
  * Delivery innovation: Yogurt matrix protects probiotics against surgical gut pH changes.
  Other Names: Maltodextrin + Guar Gum + L. rhamnosus GG; Prebiotic + Probiotic Blend; PHGG + LGG
  Arms: Intervention Group (Probiotic and Prebiotic)

SUMMARY:
This randomized controlled clinical study investigates the effects of daily synbiotic supplementation (containing Lactobacillus rhamnosus GG and partially hydrolyzed guar gum) in patients who underwent sleeve gastrectomy. 60 participants aged 18-65 with a BMI of 35 or higher were randomly assigned to intervention (n=30) and control (n=30) groups. The intervention group received a 5 g sachet daily for 12 weeks postoperatively, mixed into 200 ml of yogurt and consumed during afternoon snacks. The control group received no supplementation. Anthropometric measurements, biochemical parameters, and gastrointestinal outcomes were assessed at baseline, week 4, and week 12. The aim is to evaluate the influence of probiotic and prebiotic supplementation on gastrointestinal function and biochemical markers in the early postoperative period following bariatric surgery.

DETAILED DESCRIPTION:
Obesity is a growing global health problem, and bariatric surgery particularly sleeve gastrectomy, has become an effective method for long-term weight management. However, postoperative gastrointestinal changes, dysbiosis, and metabolic adaptations remain significant challenges, especially during the initial recovery period. The gut microbiota plays a critical role in digestion, nutrient absorption, immune modulation, and metabolic regulation. Probiotics and prebiotics may contribute to restoring microbial balance, enhancing intestinal barrier integrity, and improving biochemical profiles following surgery.

This randomized controlled trial was designed to evaluate the impact of synbiotic supplementation on gastrointestinal symptoms and selected biochemical parameters in patients undergoing sleeve gastrectomy. A total of 60 patients aged 18 to 65 years, with a body mass index (BMI) of 35 or higher, were enrolled. Participants were randomly assigned to two groups in a 1:1 ratio. The intervention group (n = 30) received a 5 g sachet containing maltodextrin (4.9 g) and Lactobacillus rhamnosus GG (1×10⁹ CFU) in a partially hydrolyzed guar gum matrix, administered once daily mixed into 200 ml of yogurt for 12 weeks postoperatively. The control group (n = 30) received no supplementation.

In the early postoperative period, patients commonly experience gastrointestinal symptoms such as bloating, gas, and constipation. This study aims to determine whether synbiotic supplementation can alleviate these symptoms and positively affect gastrointestinal function, anthropometric measurements, and specific biochemical markers. Additionally, it explores participants' knowledge and awareness of microbiota-related concepts, including probiotics and prebiotics. Data were collected through validated questionnaires assessing gastrointestinal symptoms, constipation severity, dietary habits, and microbiota-related knowledge. Anthropometric and biochemical assessments were conducted at baseline and at weeks 4 and 12 postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation (provided informed consent)
* Age between 18 and 65 years
* Body mass index (BMI) ≥ 35 kg/m²
* Underwent laparoscopic sleeve gastrectomy

Exclusion Criteria:

* Use of antibiotics for more than 5 days after surgery
* Antibiotic use within 6 months prior to surgery
* Use of any prebiotic or probiotic supplement within 3 months prior to surgery
* Known intolerance to prebiotics or probiotics
* Use of immunosuppressive drugs or NSAIDs
* Diagnosed with liver or kidney failure
* Age under 18 or over 65
* History of cholecystectomy or scheduled simultaneous cholecystectomy with sleeve gastrectomy
* Lactose intolerance
* Presence of early postoperative complications (e.g., bleeding, persistent vomiting, fistula, obstruction, leakage, infection, etc.)
* Diagnosed dumping syndrome after surgery
* Early postoperative food intolerance or dehydration
* Inability to undergo bioelectrical impedance analysis (e.g., pacemaker, metallic implants)
* Conditions affecting body composition analysis results, such as:
* Menstruation at the time of measurement
* Consumption of food or caffeinated beverages within 4 hours of measurement
* Intense physical activity within 48 hours of measurement
* Non-adherence to daily probiotic/prebiotic supplementation protocol during the intervention period Alcohol consumption within 48 hours of measurement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Change in Gastrointestinal Symptom Rating Scale (GSRS) Scores | Baseline, Week 4, Week 12
  The Gastrointestinal Symptom Rating Scale (GSRS) was used to evaluate participants' gastrointestinal symptoms before surgery, at 4 weeks post-surgery, and at 12 weeks post-surgery. The scale has five subscales targeting abdominal pain, reflux, diarrhea, indigestion, and constipation. Higher scores on the scale indicate more severe symptoms. Between-group comparisons were conducted using independent t-test and changes over time were analyzed with 2 (group) × 3 (time) repeated measures ANOVA.
Constipation Severity Scale (CSS) Score | Baseline, week 4, week 12
  The Constipation Severity Scale (CSS) was administered to participants before surgery, at 4 weeks post-surgery, and at 12 weeks post-surgery. It is a measure designed to determine the frequency, intensity, and difficulty/strain of bowel movements. The scale consists of 16 questions. The CCS has three subscales: Stool Impaction, Colon Sluggishness, and Pain. The score for the Stool Impaction subscale ranges from 0 to 28, the score for the Colon Sluggishness subscale ranges from 0 to 29, and the score for the Pain subscale ranges from 0 to 16. The total score that can be obtained from the CSS ranges from a minimum of 0 to a maximum of 73. A high score on the scale indicates the severity of the symptoms. Between-group comparisons were conducted using independent t-test and changes over time were analyzed with 2 (group) × 3 (time) repeated measures ANOVA.
Gas/Bloating Scale | Baseline, week 4, week 12
  The Gas/Bloating Scale was used to determine participants' gas/bloating symptoms before surgery, at 4 weeks post-surgery, and at 12 weeks post-surgery. It is designed to measure the frequency, severity, impact, and discomfort caused by gas/bloating symptoms. The scale consists of 12 questions, with each question scored on a scale from 0 to 4. According to the scoring system, 0 points indicate no symptoms, 1 point indicates minimal symptoms, 2-5 points indicate mild symptoms, 6-13 points indicate moderate symptoms, and 14 or more points indicate severe symptoms. Between-group comparisons were conducted using the chi-square and changes over time were analyzed with 2 (group) × 3 (time) repeated measures ANOVA.
Bristol Stool Consistency Scale | Baseline, week 4, week 12
  The Bristol Stool Consistency Scale is a scale of stool types ranging from the hardest to the softest. Type 1 stool is considered to be hard, nut-like lumps that are difficult to pass through the intestines. Type 2 stool is also lumpy but sausage-shaped. Types 1 and 2 are considered abnormally hard stools. Type 3 stools have cracks on the surface and are sausage-shaped, Type 4 stools are smooth and soft like a snake, and Type 5 stools are soft pieces with distinct edges and are easy to pass. Types 3, 4, and 5 are generally considered "normal" stool forms. The Friedman test was applied to evaluate the distribution of changes in Bristol scores over time in the study and control groups before surgery, at 4 weeks post-surgery, and at 12 weeks post-surgery. The chi-square test was used to compare the distribution and statistical comparisons of the study and control groups before surgery and at 4 and 12 weeks post-surgery according to the Bristol Stool Consistency Scale.
Change in Blood Glucose and Insulin Parameters | Baseline, Week 4, Week 12
  Blood glucose homeostasis was evaluated using fasting glucose (mg/dL), fasting insulin (µIU/mL), and HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) index, calculated using the formula [fasting blood sugar (mg/dL) x fasting insulin (µIU/mL)/405]. All values were extracted from clinical records at three time points. These variables were analyzed separately.An independent t-test was used to assess whether there were statistically significant differences between the groups.
Change in Lipid Biomarkers | Baseline, Week 4, Week 12
  To evaluate the participants' blood lipid profiles, the following parameters were assessed:
  Cholesterol (mg/dL), HDL (High-Density Lipoprotein) (mg/dL), LDL (Low-Density Lipoprotein) (mg/dL), Triglycerides (mg/dL). Each value was extracted from medical records and analyzed separately. Independent t-tests were used to compare values between intervention and control groups.
Change in Liver Function and Related Biochemical Parameters | Baseline, Week 4, Week 12
  Liver function and associated biomarkers were evaluated through the following laboratory values:
  Alanine Aminotransferase - ALT (U/L) Aspartate Aminotransferase - AST (U/L) Gamma-Glutamyl Transferase - GGT (U/L) Values were obtained from participants' medical records and assessed at baseline, 4th and 12th postoperative weeks. Independent t-tests were used to compare values between intervention and control groups.
Other biochemical parameters | Baseline, Week 4, Week 12
  Serum uric acid (mg/dL) Total Bilirubin (mg/dL) Direct Bilirubin (mg/dL) levels were assessed in all participants at three time points: before surgery, and at 4 and 12 weeks postoperatively. Values were obtained from patient medical records. Differences between intervention and control groups were analyzed using independent t-tests.

SECONDARY OUTCOMES:
Change in anthropometric measurements | Baseline, Week 4, Week 12
  Anthropometric data were collected at three different time points to assess changes in body composition. Body mass index (BMI) was calculated using the formula kg/m^2 based on the obtained height and body weight. At each time point (baseline, week 4, week 12), intergroup comparisons were reported using independent t-tests to identify statistically significant differences. Measurements were performed under standard conditions at each time point.
Change in Body Composition Parameters | Baseline, Week 4, Week 12
  Body composition was evaluated using a standardized protocol and the same device (Tanita MC-780, bioelectrical impedance analyzer) across all time points. The following parameters were assessed:
  Body weight (kg) Body fat mass (kg) Skeletal muscle mass (kg) Total body water (kg) All values were measured under fasting and standardized conditions. Results were analyzed individually.
Change in physical activity levels | Baseline, Week 4, Week 12
  Participants' physical activity levels were assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). Scores were calculated in weekly MET-minutes. Higher scores indicate higher activity levels. The Total Physical Activity Score (TPAS) was calculated as Walking (+) Moderate-intensity activity (+) Vigorous-intensity activity score.
  As a result, physical activity level was classified as:
  * TPAS <600 MET: 'Not physically active'
  * TPAS = 600-3000 MET is defined as 'Low Physical Activity Level'
  * TPAS ≥ 3000 MET is defined as 'Adequate Physical Activity Level' To assess differences in physical activity levels over time, independent t-tests were used at each time point to compare groups.
Baseline group differences in Microbiota Awareness Scores (MAS) | Baseline only
  Participants' awareness of concepts such as microbiota, probiotics, and prebiotics was assessed before surgery using the Microbiota Awareness Scale (MAS). The scale includes four subdomains: general knowledge, product knowledge, chronic diseases, and probiotics/prebiotics. A total awareness score was also calculated. Scores range from 18 to 100, with higher scores indicating greater awareness. Differences between the intervention and control groups were analyzed using independent t-tests. Additionally, subgroup comparisons were conducted to evaluate awareness levels across different educational backgrounds.

CONTACTS AND LOCATIONS:
Overall Officials: Ayhan Dağ, Assoc. Prof., Study Chair — Lokman Hekim University
Locations (1):
- Türk Obezite Cerrahisi Vakfı, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This is a graduate thesis project. Individual participant data will not be shared. The data is stored securely and used solely for academic research, as approved by the ethics committee.